CLINICAL TRIAL: NCT01965925
Title: Targeting Circadian and Cognitive Dysfunction in Bipolar Disorder With Modafinil
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Katherine Burdick, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 12-1573; R34MH101267 (NIH)
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Bipolar Disorder
Keywords: Cognition; Sleep problems; Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder; Parasomnias | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modafinil (Experimental): Modafinil will be administered at baseline with a single dose of 100 mg/day QAM increased at week 1 to a single dose 200mg/day QAM. Patients will take drug upon waking with no adjustment in sleep schedule. Dosing will be flexible based on side effects with a maximum dose of 200 mg/day. Subjects will be discontinued if 100mg/day is not tolerated.
  Interventions: Drug: Modafinil
- Placebo (Placebo Comparator): Subjects will take placebo upon waking once per day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modafinil — Ratio of 2:1 subjects will be in the experimental arm receiving modafinil for 8 weeks.
  Arms: Modafinil
Drug: Placebo — For every randomly assigned 2 subjects receiving active drug, 1 will be randomly assigned to receive placebo for 8 weeks.
  Arms: Placebo

SUMMARY:
This is an 8-week, randomized, placebo-controlled trial of modafinil in stable bipolar disorder patients. Results will provide information on a promising treatment for simultaneously treating both sleep and cognitive problems in stable bipolar patients. These disabling symptoms persist despite stable mood and are strongly associated with functional disability, making them important treatment targets that have not yet been adequately addressed.

DETAILED DESCRIPTION:
Changes in the sleep-wake cycle are other circadian rhythms represent core features of Bipolar Disorder (BD), with sleep abnormalities in approximately 90% of patients during acute episodes. Even when euthymic, many BD patients continue to demonstrate circadian disruptions, including diminished sleep efficiency and lower daytime activity levels (Plante, 2008). Moreover, unaffected offspring of BD patients demonstrate sleep and activity abnormalities (Ankers, 2009), and variation within several circadian-related genes (e.g. CLOCK) has been associated with risk for BD (Dallaspezia, 2009). These trait-like circadian disruptions are of particular clinical relevance as chances in sleep are highly predictive of impending affective instability (Plante, 2008) and BD patients with poor sleep quality report diminished quality of life (Gruber, 2009). Psychosocial treatments that incorporate the regulation of sleep and activity in BD have been successful in reducing recurrence, highlighting the important of stabilizing circadian rhythms in BD (Frank, 2005); yet treatment remains suboptimal and, to date, no pharmacological intervention using circadian measures as outcomes in BD has been published.

The exact nature of the circadian abnormality in BD is known; theories posit a potential uncoupling of the biological clock from external variables that entrain circadian rhythms (e.g. light) versus the desynchronization of the sleep-wake cycle such that it falls out of phase with other biological rhythms (Dallaspezia, 2009). Euthymic BD patients are commonly characterized by an eveningness chronotype, such that their time-to-sleep preference is phase-shifted to a later than average hour, one that is not typically aligned with the 24-hour light-dark cycle (Plante, 2008; Ahn, 2008). Potential consequences related to these persistent circadian abnormalities include significant reductions in daytime wakefulness and neurocognitive impairment.

While sleep deprivation induced by single-trial phase-shifts only impairs cognition until sleep in recovered, chronic deprivation such as those noted in BD individuals, have been implicated in significant learning and memory deficits in animal models (Craig, 2008). Moreover, humans who are unable to synchronize normal sleep-wakefulness schedules with their own internal biological clocks are impaired on tasks of processing speed, working memory, and learning (Wright, 2006). Indeed, a majority of BD patients demonstrate deficits in attention, memory, and executive function even when affectively stable (Goldberg & Burdick, 2008). Although several features of the illness potentially contribute to the persistent cognitive impairment noted during euthymic periods, the circadian-based deficits in sleep quality and daytime wakefulness are likely to exacerbate cognitive problems in BD (Giglio, 2010), as has been shown in healthy controls, sleep disordered subjects and other clinical conditions (Benca, 2009). Preliminary data support this relationship in BD. The possible influence of chronic circadian disruption on cognition in BD is of critical importance because of a strong association between cognition during euthymic and functional disability (Sanchez-Moreno, 2009).

When considering agents that may simultaneously improve upon sleep quality and enhance cognition, the wake-promoting agents, modafinil, is an ideal candidate. It is FDA approved for improving wakefulness in adults with excessive daytime sleepiness due to primary sleep disorders (Provigil, 2007) and is characterized as a psychostimulant but has been differentiated from amphetamine by a lower liability for abuse and a more favorable risk profile. Modafinil has been shown to enhance cognition in healthy controls, sleep-disordered individuals, neurological patients, and patients with schizophrenia (Minzenberg, 2008). Preliminary data indicate that modafinil is safe and effective as an adjunctive in depressed BD patients, with no risk for mania-induction vs placebo (Frye, 2007); however there has not yet been a systematic trial in euthymic BD patients with sleep and cognitive dysfunction as outcome measures. Thus, adjunctive modafinil (200 mg/day) vs placebo will be administered to 48 euthymic patients with BD for 8 weeks with three specific aims:

1. To evaluate the safety of adjunctive modafinil in euthymic BD. Adverse events will be carefully measured and recorded in an effort to determine the base rates for common side effects in BD. Specifically, mood and psychosis ratings will be conducted weekly to address the potential for modafinil to exacerbate manic and/or psychotic symptoms.
2. To evaluate the effects of adjunctive modafinil in euthymic BD on measures of sleep quality and daytime wakefulness. Patients' subjective experience of sleep disruption and daytime wakefulness will be measured weekly using several standard questionnaires and daily diaries.
3. To evaluate the effects of adjunctive modafinil in euthymic BD on measures of neurocognition. Cognitive functioning will be assayed using the MATRICS Consensus Cognitive Battery supplemented by several domain-specific tasks at baseline, 4-weeks, and at the end of the 8-week study.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV Bipolar Disorder I or Bipolar Disorder II diagnosis
* Affectively stable
* Clinically acceptable, stably-dosed, mood stabilizing medication regimen for > 1 month prior to enrollment, with no medication changes planned over the 8-week study period.
* Objective evidence of either a subjective sleep quality complaint and/or clinically-significant cognitive impairment at screening.

Exclusion Criteria:

* History of Central Nervous System trauma, neurological disorder, ADHD, or a learning disability.
* Positive urine toxicology or DSM-IV diagnosis of substance abuse/dependence within 3 months
* Active, unstable medical problem that may interfere with sleep and/or cognition.
* History of substance induced mania
* Recent history of rapid cycling
* Score of 2 or greater on the decreased need for sleep item on CARS-M
* Any drug known to interfere with modafinil
* More than 2 psychotropic medications
* Abnormal lab or ECG result at screen
* Significant suicidal ideation at baseline or at risk for suicidal behavior based on clinical judgment
* participation in any other investigational cognitive enhancement study within 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-01; Primary Completion 2017-11-09 (Actual); Study Completion 2017-11-09 (Actual)

PRIMARY OUTCOMES:
safety of adjunctive modafinil | up to 8 weeks
  Adverse events will be carefully measured and recorded in an effort to determine the base rates for common side effects in BD. Specifically, mood and psychosis ratings will be conducted.

SECONDARY OUTCOMES:
MCCB | baseline
  MATRICS Cognitive Consensus Batter to assess cognitive functioning
MCCB | week 4
  MATRICS Cognitive Consensus Batter to assess cognitive functioning
MCCB | week 8
  MATRICS Cognitive Consensus Batter to assess cognitive functioning
sleep quality | baseline
  To evaluate the effects of adjunctive modafinil in euthymic BD on measures of sleep quality and daytime wakefulness, using Pittsburgh Sleep Quality Index (PSQI) and Epworth Sleepiness Scale (ESS)
sleep quality | week 4
  To evaluate the effects of adjunctive modafinil in euthymic BD on measures of sleep quality and daytime wakefulness, using Pittsburgh Sleep Quality Index (PSQI) and Epworth Sleepiness Scale (ESS)
sleep quality | week 8
  To evaluate the effects of adjunctive modafinil in euthymic BD on measures of sleep quality and daytime wakefulness, using Pittsburgh Sleep Quality Index (PSQI) and Epworth Sleepiness Scale (ESS)
UPSA | baseline
  UCSC Performance Skills Assessment assess functional ability
UPSA | week 4
  UCSC Performance Skills Assessment assess functional ability
UPSA | week 8
  UCSC Performance Skills Assessment assess functional ability
QoL | baseline
  Quality of Life Scale
QoL | week 4
  Quality of Life Scale
QoL | week 8
  Quality of Life Scale
Vital signs | up to 8 weeks
  vital signs including blood pressure
Electrocardiogram | baseline and week 8
  comparison of electrocardiogram (EKG) results from week 8 to baseline.
liver function tests | baseline and week 8
  comparison of liver function test results from week 8 to baseline
chemistry panel | baseline and week 8
  comparison of chemistry panel results from week 8 to baseline
Complete blood count | baseline and week 8
  comparison of complete blood count (CBC) results from week 8 to baseline
urinalysis | baseline and week 8
  comparison of urinalysis results from week 8 to baseline
Suicide risk scale | up to 8 weeks
  Beck Scale for Suicidal Ideation and Columbia Suicide Severity Rating Scales
Medication log | up to 8 weeks
  Medication log for current medications and all medications administered

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Burdick, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Lipschitz JM, Perez-Rodriguez M, Majd M, Larsen E, Locascio J, Pike CK, Shanahan M, Burdick KE. Modafinil's effects on cognition and sleep quality in affectively-stable patients with bipolar disorder: a pilot study. Front Psychiatry. 2023 Sep 4;14:1246149. doi: 10.3389/fpsyt.2023.1246149. eCollection 2023. PMID 37732080